CLINICAL TRIAL: NCT00233233
Title: Assessment Mode and Validity of Self-Reports in Adults
Brief Title: Influence of Data Collection Mode on Self-Report Validity of Asthma Therapy Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized
Other Study IDs: 325; R01HL064200 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Lung Diseases; Asthma
MeSH Terms: conditions — Lung Diseases; Asthma

INTERVENTIONS:
Behavioral: Standardized Asthma Education Program

SUMMARY:
This study will examine how the assessment mode influences the validity of self-reported adherence to asthma therapy. Self-reported adherence to asthma therapy data will be collected using one of three randomized assessment modes (interview, computer, or telephone).

DETAILED DESCRIPTION:
BACKGROUND:

Self-reports are a primary source of behavioral data. Studies have highlighted the variable validity and reliability of self-report measures of health behaviors such as adherence to therapy. Research on self-reports of sensitive information, such as sexual behavior and drug use, suggests that the mode of data collection may enhance validity of self-reports. However, no studies have determined how the mode of data collection influences self-reports when an objective measure of the behavior is available.

DESIGN NARRATIVE:

The primary aim of this study is to examine the influence of the mode of data collection on the validity of self-reports of inhaled anti-inflammatory medication adherence.

The key secondary outcomes of the study will attempt to answer the following questions: 1) does the assessment mode influence self-reports of commonly used asthma outcome measures of disease-related symptoms, self-management behaviors, and quality of life?; 2) does the relationship between the assessment mode, the validity of self-reports of adherence, and other measures (i.e., asthma symptoms, self-management behaviors, and quality of life) change over time?; and 3) does the assessment mode interact with baseline personality characteristics and mood to influence the validity of self-reports of adherence and other outcome measures (i.e., asthma symptoms, self-management behaviors, and quality of life)?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Under a provider's care for asthma
* Prescribed daily inhaled corticosteroids (by metered dose inhaler [MDI]) at least 2 times a day
* Speaks English
* Otherwise in good general health

Exclusion Criteria:

N/A

Ages: 19 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2002-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Concordance between patient's self-reported medication adherence and electronically measured adherence | Measured at Months 1 through 5

SECONDARY OUTCOMES:
Impact of mode of assessment on adult self-reports of asthma symptoms, asthma management practices, and quality of life | Measured at Months 1 through 5
Relationship between baseline measures of psychosocial variables (i.e., personality and mood) and the primary outcome | Measured at Months 1 through 5

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Rand, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States